CLINICAL TRIAL: NCT07404501
Title: A Gamified Approach To Burn Education And Prevention Among Youth: The Randomized Controlled Study "Burn Game"
Brief Title: Gamified Approach To Burn Education - Randomized Controlled Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 90231725.9.0000.0068
Record Dates: First submitted 2026-02-04; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Burn; Health Education; Accident Prevention; First Aid; Educational Intervention; Game-based Education
Keywords: Burns; Health Education; Accident Prevention; First Aid; Educational Games
MeSH Terms: conditions — Burns; Health Education | interventions — First Aid

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Serious Digital Game (Experimental): Participants in this arm will receive a brief standardized introductory session covering basic concepts of burns, including causes, prevention, and first aid. After this introduction, participants will engage in a serious digital game for 25 minutes following a 5-minute familiarization period with the platform, totaling 30 minutes. The game presents educational content and questions related to burn prevention and first aid through virtual avatars. Participants are required to consult in-game educational materials before answering questions. Performance is assessed based on accuracy and response time, generating an automated final score. Participants will complete a post-intervention knowledge assessment questionnaire and a satisfaction questionnaire at the end of the intervention, as well as a follow-up assessment two weeks later.
  Interventions: Behavioral: Serious Digital Game for Burn Prevention and First Aid
- Face-to-Face Educational Lecture (Active Comparator): Participants in this arm will first receive a brief standardized introductory session covering basic concepts of burns, including causes, prevention, and first aid. After this introduction, participants will attend a face-to-face educational lecture lasting 30 minutes, addressing types of burns, etiology, prevention strategies, and basic first-aid measures. Participants will complete pre- and post-intervention knowledge assessment questionnaires, as well as a follow-up assessment two weeks after the intervention.
  Interventions: Behavioral: Face-to-Face Educational Lecture on Burn Prevention and First Aid

INTERVENTIONS:
Behavioral: Serious Digital Game for Burn Prevention and First Aid — The intervention consists of a serious digital game designed to provide education on burn prevention and first aid. The game delivers educational content through an interactive virtual environment in which participants engage with avatars that present questions and learning challenges related to burns. Participants are required to consult in-game educational materials before responding to each question. Performance metrics, including response accuracy and time to answer, are recorded automatically by the system to generate an overall score - which is not an endpoint of this study, since the control group does not have access to the game. The intervention is intended to promote active learning and knowledge acquisition through interactive and gamified educational strategies.
  Arms: Serious Digital Game
Behavioral: Face-to-Face Educational Lecture on Burn Prevention and First Aid — The intervention consists of an in-person 30-minute educational lecture focused on burn prevention and first aid. The lecture is designed to deliver structured educational content in a didactic format, covering key topics related to burns, including common causes, prevention strategies, and basic first-aid measures. The session is conducted by a trained instructor and aims to provide participants with foundational knowledge through direct instruction, without the use of interactive gaming components.
  Arms: Face-to-Face Educational Lecture

SUMMARY:
The goal of this clinical trial is to evaluate whether different educational strategies can improve knowledge acquisition regarding burn prevention and first aid among students enrolled in a community-based preparatory course. The main questions it aims to answer are:

Does participation in a serious digital game improve knowledge about burn prevention and first aid compared with a traditional lecture? Researchers will compare a serious digital game with a face-to-face educational lecture to determine differences in knowledge acquisition and participant satisfaction between the two educational approaches.

Participants will:

Receive a brief (5 minutes) standardized introductory explanation about basic concepts of burns; Be randomized to participate in either a serious digital game or a face-to-face educational lecture; Complete knowledge assessment questionnaires prior to and after the intervention; Complete a satisfaction questionnaire; Attend a follow-up assessment two weeks after the intervention.

DETAILED DESCRIPTION:
This study is a randomized, single-blind, behavioral and educational intervention with two parallel arms designed to evaluate different educational strategies for burn prevention and first aid.

All participants will initially receive a brief (5 minutes) standardized introductory session covering basic concepts related to burns, including definition, common causes, prevention strategies, and first-aid measures. This introductory explanation is intended to ensure that all participants have a minimum and uniform baseline understanding of the topic prior to the intervention.

After this initial session, participants will be randomly allocated to one of two intervention groups.

Participants allocated to the serious digital game group will receive a 5-minute familiarization period with the digital platform, followed by 25 minutes of gameplay. The serious game presents educational content and questions related to burn prevention and first aid through virtual avatars, requiring participants to consult in-game educational materials before answering questions. Performance is recorded automatically by the game system.

Participants allocated to the face-to-face educational lecture group will attend an in-person lecture lasting approximately 30 minutes. The lecture will address types of burns, etiology, prevention measures, and basic first-aid management in primary health care.

Knowledge acquisition will be assessed using structured multiple-choice questionnaires administered prior to and after the intervention. Participant satisfaction will also be evaluated using a Likert-scale questionnaire. A follow-up assessment will be conducted two weeks after the intervention to evaluate knowledge retention.

Outcome assessment will be performed by an evaluator blinded to group allocation. Sociodemographic variables, including age, sex, and socioeconomic status, will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Students regularly enrolled in the MedEnsina preparatory course
* Ability to understand the instructions and the content of the proposed educational activities
* Availability to participate in the intervention on the first day of the study and to attend the two-week follow-up
* Signed informed consent form and, when applicable, assent form

Exclusion Criteria:

* Failure to attend the intervention on the first day of the study
* Failure to attend the follow-up assessment two weeks after the intervention
* Incomplete completion of the pre- or post-intervention questionnaires
* Withdrawal of consent at any stage of the study
* Any condition that, in the investigators' judgment, may impair adequate participation or understanding of the educational activities

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Change in Knowledge Scores on Burn Prevention and First Aid After the Educational Interventions | From baseline to immediately post-intervention
  The primary outcome is knowledge acquisition related to burn prevention and first aid. Knowledge will be measured using a structured multiple-choice questionnaire administered immediately before and immediately after the educational intervention. The questionnaire consists of 20 questions covering basic concepts of burns, prevention strategies, and first-aid measures. Each correct answer contributes to the total knowledge score, with higher scores indicating greater knowledge. The primary outcome will be expressed as the change in knowledge score from baseline to immediately after the intervention and compared between the two educational groups.

SECONDARY OUTCOMES:
Knowledge Retention Scores After the Educational Interventions | From baseline to 2 weeks post-intervention
  Knowledge retention related to burn prevention and first aid will be assessed using the same structured multiple-choice questionnaire applied during the initial evaluation. The 20-question questionnaire will be administered again approximately two weeks after the educational intervention to evaluate how much of the information learned was retained over time. The total score obtained at the follow-up assessment will be compared with the baseline and immediate post-intervention scores. Higher scores indicate greater retention of knowledge.

OTHER OUTCOMES:
Participant Satisfaction With the Educational Interventions | Immediately after the intervention
  Participant satisfaction with the educational intervention will be assessed immediately after completion of the intervention. Satisfaction will be measured using a structured questionnaire based on a Likert scale (USERQ), validated for Brazilian Portuguese. The questionnaire evaluates participants' perceptions of the educational experience, including clarity of content, engagement, usability, and overall satisfaction. Higher scores indicate greater participant satisfaction with the educational intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Pires Camargo, Md, PhD, Principal Investigator — Laboratory of Plastic Surgery and Regenerative Medicine, School of Medicine, Universidade de São Paulo, SP, Brazil
Locations (1):
- School of Medicine, Universidade de São Paulo, SP, Brazil, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared because the study involves educational interventions with students and includes potentially sensitive personal and sociodemographic information. Data sharing was not included in the ethics committee approval, and participant consent did not authorize public sharing of individual-level data. Only aggregated and anonymized results will be reported.